CLINICAL TRIAL: NCT05578248
Title: The Andrews Return to Sport ACL Score: A Developmental Study
Brief Title: Andrews Return to Sport ACL Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Return to Sport
Record Dates: First submitted 2022-09-30; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: ACL Injury
Keywords: Cohort; return to sport
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Collegiate Athletes: Group designated for collegiate athletes; see protocol for treatment plan
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Procedure: ACL reconstruction
- Pre-collegiate Athletes: Group designated for pre-collegiate, or high school-age, athletes; see protocol for treatment plan
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Procedure: ACL reconstruction

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Non-invasive imaging technology that produces three-dimensional detailed anatomical images
Procedure: ACL reconstruction — Surgical procedure to repair damaged or severed anterior cruciate ligament in the knee

SUMMARY:
This project will develop a data-driven decision making model to assess a competitive athlete's readiness to return to sport after ACL injury and surgery safely.

DETAILED DESCRIPTION:
One hundred pre-collegiate or collegiate athlete participants will be recruited for this study. The duration of the treatment plan will be 24 months. Each of the participants will be qualified for the study due to falling within all inclusion criterion and no exclusion criterion. The screening of the inclusion criterion will occur at visit one of the study. At this time, the AREF Research Team will review and collect informed consent from each participant. Visit two will occur three (3) months after each participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician will occur along with functional movement assessment and MRI. Visit three will occur six (6) months after each participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician will occur along with functional movement assessment and MRI. Visit four will occur nine (9) months after each participant's ACL reconstruction surgery. At this time, an medical evaluation by the treating leading physician will occur along with functional movement assessment and MRI. Visit five will occur twelve (12) months after each participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician will occur along with functional movement assessment and MRI. Visit six will occur eighteen (18) months after each participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician will occur along with functional movement assessment and MRI. Visit seven will occur twenty-four (24) months after each participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician will occur along with functional movement assessment and MRI. At each time point, the treating physician or the therapist performing the functional movement assessment can choose to limit the functional movement assessment if there are concerns that the patient may not be ready for the expected load of one or more elements of the functional movement assessment.

At each monthly time point after ACL reconstruction, patient reported outcomes will be collected by the research team to assist in assessing the overall health and confidence in return to sport for each athlete. The following patient reported outcomes will be collected in written or electronic format after informed consent has been obtained from each participant: Sports Participation, Reinjury, Tampa Kinesiophobia Scale, IKDC, PROMIS, SANE.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-24 years
* Require ACL reconstruction surgery
* No other ligament injury which would require repair or reconstruction to lower extremity is present as assessed by treating physician
* Exhibits desire to return to pre-injury competitive level
* Assessed to be in good physical health condition by the treating physician

Exclusion Criteria:

* Requires more than one ACL reconstruction surgery at time of screening
* Has comorbid lower extremity diagnoses which would impede return to sport as assessed by the treating physician
* Does not desire to return to pre-injury competitive sport level

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 competitive pre-collegiate or collegiate athletes who have recently suffered from an ACL injury that requires reconstructive surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia | Through study completion, an average of 1 year
  Measurement to determine the physical and pyschological effects on the rehabilitation of an injured athlete; 17-question survey with a total score calculated after inversion of the individual scores of items 4, 8, 12, and 16 (all questions are scored on a scale of 1-4 points).
Sports Participation Assessment | Through study completion, an average of 1 year
  Quantifies the participant's participation in sports activity during the rehabilitation period
Reinjury Assessment | Through study completion, an average of 1 year
  Monthly questionnaire to assess the rate of reinjury during rehabilitation process
International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) | Every month, up to 1 year; assessing for change
  19-question form that will contribute to comprehensive data set by evaluating confidence in perfomance
Patient Reported Outcomes Measurement Information Systems (PROMIS) | Every month, up to 1 year; assessing for change
  Assesses overall health functioning and rehabilitation levels of each participant; required to ensure that a comprehensive assessment of overall functioning is reviewed. Scores range from 20 to 80, with 50 representing the average for the general population, and increases in this number over 50 represent standard deviation, and thus represent slow recovery progress in this study
Single Assessment Numeric Evaluation (SANE) | Every month, up to 1 year; assessing for change
  Single question PRO with a rating of 0-100 for each participant to score their current functioning in comparison to their pre-injury level of function

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Andrews Research and Education Foundation, Gulf Breeze, Florida, United States

REFERENCES:
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br J Sports Med. 2014 Nov;48(21):1543-52. doi: 10.1136/bjsports-2013-093398. Epub 2014 Aug 25. PMID 25157180
- [Background] Bodor M. Quadriceps protects the anterior cruciate ligament. J Orthop Res. 2001 Jul;19(4):629-33. doi: 10.1016/S0736-0266(01)00050-X. PMID 11518272
- [Background] Brodke DJ, Saltzman CL, Brodke DS. PROMIS for Orthopaedic Outcomes Measurement. J Am Acad Orthop Surg. 2016 Nov;24(11):744-749. doi: 10.5435/JAAOS-D-15-00404. PMID 27661391
- [Background] Boyle, M. & Galway, B.(n.d.). Evidence-based Clinical Protocols: Anterior Cruciate Ligament Injury & Reconstruction. Biodex Medical Systems, Inc.
- [Background] Creighton DW, Shrier I, Shultz R, Meeuwisse WH, Matheson GO. Return-to-play in sport: a decision-based model. Clin J Sport Med. 2010 Sep;20(5):379-85. doi: 10.1097/JSM.0b013e3181f3c0fe. PMID 20818198
- [Background] Davies GJ, McCarty E, Provencher M, Manske RC. ACL Return to Sport Guidelines and Criteria. Curr Rev Musculoskelet Med. 2017 Sep;10(3):307-314. doi: 10.1007/s12178-017-9420-9. PMID 28702921
- [Background] Gianotti SM, Marshall SW, Hume PA, Bunt L. Incidence of anterior cruciate ligament injury and other knee ligament injuries: a national population-based study. J Sci Med Sport. 2009 Nov;12(6):622-7. doi: 10.1016/j.jsams.2008.07.005. Epub 2008 Oct 2. PMID 18835221
- [Background] Griffin LY, Agel J, Albohm MJ, Arendt EA, Dick RW, Garrett WE, Garrick JG, Hewett TE, Huston L, Ireland ML, Johnson RJ, Kibler WB, Lephart S, Lewis JL, Lindenfeld TN, Mandelbaum BR, Marchak P, Teitz CC, Wojtys EM. Noncontact anterior cruciate ligament injuries: risk factors and prevention strategies. J Am Acad Orthop Surg. 2000 May-Jun;8(3):141-50. doi: 10.5435/00124635-200005000-00001. PMID 10874221
- [Background] Grindem H, Snyder-Mackler L, Moksnes H, Engebretsen L, Risberg MA. Simple decision rules can reduce reinjury risk by 84% after ACL reconstruction: the Delaware-Oslo ACL cohort study. Br J Sports Med. 2016 Jul;50(13):804-8. doi: 10.1136/bjsports-2016-096031. Epub 2016 May 9. PMID 27162233
- [Background] Gokeler A, Welling W, Zaffagnini S, Seil R, Padua D. Development of a test battery to enhance safe return to sports after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2017 Jan;25(1):192-199. doi: 10.1007/s00167-016-4246-3. Epub 2016 Jul 16. PMID 27423208
- [Background] Jordan MJ, Morris N, Lane M, Barnert J, MacGregor K, Heard M, Robinson S, Herzog W. Monitoring the Return to Sport Transition After ACL Injury: An Alpine Ski Racing Case Study. Front Sports Act Living. 2020 Mar 3;2:12. doi: 10.3389/fspor.2020.00012. eCollection 2020. PMID 33345007
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Lundberg M, Styf J, Jansson B. On what patients does the Tampa Scale for Kinesiophobia fit? Physiother Theory Pract. 2009 Oct;25(7):495-506. doi: 10.3109/09593980802662160. PMID 19925172
- [Background] Manske R, Reiman M. Functional performance testing for power and return to sports. Sports Health. 2013 May;5(3):244-50. doi: 10.1177/1941738113479925. PMID 24427396
- [Background] Miller RP, Kori S, Todd D. The Tampa Scale: a measure of kinesiophobia. Clin J Pain. 1991;7(1):51-52.
- [Background] O'Connor CM, Ring D. Correlation of Single Assessment Numeric Evaluation (SANE) with other Patient Reported Outcome Measures (PROMs). Arch Bone Jt Surg. 2019 Jul;7(4):303-306. PMID 31448305
- [Background] Wilk KE, Macrina LC, Cain EL, Dugas JR, Andrews JR. Recent advances in the rehabilitation of anterior cruciate ligament injuries. J Orthop Sports Phys Ther. 2012 Mar;42(3):153-71. doi: 10.2519/jospt.2012.3741. Epub 2012 Feb 29. PMID 22382825

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05578248/Prot_000.pdf
  • Informed Consent Form (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05578248/ICF_001.pdf